CLINICAL TRIAL: NCT04726839
Title: Biomarkers algOrithm for strOke diagnoSis and Treatment Resistance Prediction
Acronym: BOOST
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200188
Record Dates: First submitted 2021-01-24; First posted 2021-01-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Ischemic; Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stroke suspicion: Patients with stroke suspicion within 24 hours of stroke's symptoms
  Interventions: Other: Standard of care for stroke management and evaluation of functionnal outcome at 3 months

INTERVENTIONS:
Other: Standard of care for stroke management and evaluation of functionnal outcome at 3 months — Additional tubes at inclusion (maximum 13 mL) Collection of the mRS data during a routine visit if planned at 3 months +/-15 days or, if not during a specific research phone call at 3 months

SUMMARY:
Triage of acute ischemic stroke (AIS) patients is critical, to decrease time to treatment, and improve functional outcome. The therapeutic standard of care for AIS consecutive to large vessel occlusion (LVO) is the association of intravenous (IV) alteplase administration and mechanical thrombectomy (MT). However, there are limited places where MT can be performed. Therefore, there is a need for innovative tools to identify, in the ambulance, patients with LVO that require MT. Sending the patients at the right, avoiding futile stops (i.e. in places where MT is not available), is definitively a strategy that saves time.

There is currently no biomarker nor Point Of Care (POC) Lab Testing to solve this issue and clinical scoring methods such as the NIHSS have a low accuracy rate to detect LVO. The relevance of blood biomarkers for LVO diagnosis and therapeutic decisions needs to be confirmed for effective triage in the setting of AIS with LVO, which represent 30% of all AIS.

The main objective of our study is to determine diagnostic performances of a panel of selected blood biomarkers to identify patients with AIS consecutive to LVO among those with stroke suspicion, within 24 hours of stroke symptom's onset before brain imaging.

This could facilitate the triage of patients with LVO refractory to thrombolysis treatment, who may benefit most from MT.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms consistent with stroke <24 hours
* Adult patients ≥ 18 years old
* Non opposition of the patient or his/her relatives to the research (emergency inclusion procedure)

Exclusion Criteria:

* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke suspicion within 24 hours of stroke's symptoms
Sampling Method: Non-Probability Sample
Enrollment: 3880 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis by the selected panel of blood biomarkers of the LVO presence eligible for MT | within 24 hours following inclusion

SECONDARY OUTCOMES:
Discrimination by the selected panel of blood biomarkers of LVO from small strokes, and AIS from hemorrhagic strokes and stroke mimics | within 24 hours following inclusion
reperfusion therapy resistance (i.e. IV thrombolysis, MT) | within 24 hours following inclusion
cardio-embolic origin | at 3 months
Early neurological improvement | at day 1 after inclusion
  Early neurological improvement will be assessed by NIHSS. Early neurological improvement will be defined as decrease of 8 points in the NIHSS or a NIHSS 0-1 within 24h for LVO confirmed patients
Functional outcome | at day 90 after inclusion
  Functional outcome will be assessed by modified Rankin Scale (mRS); It consists of a single item, with 6 levels of disability. 0 corresponding to no disability, and five to severe disability.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Department Neurology Caen Hospital, Caen
  - Lariboisière, Paris
  - Rothschild Foundation Hospital, Paris
  - Hospital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Undecided